CLINICAL TRIAL: NCT06428604
Title: The Effect of Preoperative Oral Carbohydrate Administration on Perioperative Hypothermia in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Sevil Azazoglu ERBEK, anesthesiologist, Başakşehir Çam & Sakura City Hospital
Other Study IDs: 2019/64
Record Dates: First submitted 2024-05-15; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Perioperative Hypothermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GRUP W: patient group given only 5 ml kg-1 oral water 3 hours before the surgery,
- GRUP C: Patient group given 5 ml kg-1 clear carbohydrate-rich liquid orally 3 hours before surgery

SUMMARY:
Hypothermia that may develop in the perioperative period is associated with many adverse clinical outcomes. In particular, pediatric patients were more susceptible to hypothermia and related complications such as respiratory distress, metabolic acidosis, hypoglycemia, hypoxemia, cardiac disorders, coagulopathy, and wound infection than adults. In this study, the effect of preoperative carbohydrate-rich feeding on temperature regulation in pediatric patients was investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients to be operated on by the Department of Pediatric Surgery
2. Being between the ages of 2 and 15
3. Not restricting oral intake
4. ASA I-II-III patients in anesthesia risk score
5. Patients operated between 01.03.2019 and 31.07.2019
6. Not having any communication problems (mental retardation, not knowing Turkish, etc.)
7. Not having gastroesophageal reflux
8. Not having any muscle disease
9. Informed volunteer consent must be obtained
10. Patients for whom emergency surgery is not planned
11. No disease related to the central nervous system

Exclusion Criteria:

1. Pediatric patients outside the 2-15 age range
2. Having limited oral intake
3. ASA IV and above in anesthesia risk scoring
4. Patients operated before 01.03.2019 or after 31.07.2019
5. Patients who may have communication problems with their parents or themselves
6. Patients with gastroesophageal reflux
7. Patients with muscle disease
8. Patients for whom informed voluntary consent has not been obtained
9. Patients who will undergo emergency surgery
10. Patients with diseases related to the central nervous system

Ages: 2 Years to 15 Years | Sex: All
Age Groups: Child
Study Population: Being between the ages of 2 and 15
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
the effect of oral clear liquid intake containing carbohydrates 3 hours before preoperatively on body temperature in the pediatric age group, compared to the group taking water 3 hours before surgery. | 1 March 2019- 31 july 2019
  In order to benefit from the thermic effects of nutrients, intravenous or oral administration of nutrients before or during the operation has been used. These include administering amino acid solutions and administering carbohydrate solutions Providing essential nutrients increases metabolic heat production, reducing the inequality between heat production and loss. The primary goal of this approach is to increase energy expenditure following the administration of essential nutrients, causing a response known as diet-induced thermogenesis.
  The body temperatures of the patients were measured perioperative with a tympanic thermometer at regular intervals. Values lower than 36.0oC were considered as hypothermia.

CONTACTS AND LOCATIONS:
Locations (1):
- Başakşehir Çam and Sakura City Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Yatabe T, Kawano T, Yamashita K, Yokoyama M. Preoperative carbohydrate-rich beverage reduces hypothermia during general anesthesia in rats. J Anesth. 2011 Aug;25(4):558-62. doi: 10.1007/s00540-011-1170-z. Epub 2011 May 24. PMID 21607766
- [Background] Dilmen OK, Yentur E, Tunali Y, Balci H, Bahar M. Does preoperative oral carbohydrate treatment reduce the postoperative surgical stress response in lumbar disc surgery? Clin Neurol Neurosurg. 2017 Feb;153:82-86. doi: 10.1016/j.clineuro.2016.12.016. Epub 2016 Dec 29. PMID 28073036
- [Background] Castillo-Zamora C, Castillo-Peralta LA, Nava-Ocampo AA. Randomized trial comparing overnight preoperative fasting period Vs oral administration of apple juice at 06:00-06:30 am in pediatric orthopedic surgical patients. Paediatr Anaesth. 2005 Aug;15(8):638-42. doi: 10.1111/j.1460-9592.2005.01517.x. PMID 16033337
- [Background] Carvalho CALB, Carvalho AA, Nogueira PLB, Aguilar-Nascimento JE. CHANGING PARADIGMS IN PREOPERATIVE FASTING: RESULTS OF A JOINT EFFORT IN PEDIATRIC SURGERY. Arq Bras Cir Dig. 2017 Jan-Mar;30(1):7-10. doi: 10.1590/0102-6720201700010003. PMID 28489159
- [Background] Ozer AB, Demirel I, Kavak BS, Gurbuz O, Unlu S, Bayar MK, Erhan OL. Effects of preoperative oral carbohydrate solution intake on thermoregulation. Med Sci Monit. 2013 Jul 31;19:625-30. doi: 10.12659/MSM.883991. PMID 23900128